CLINICAL TRIAL: NCT00953992
Title: The Study of Etiology, Epidemiology and Prognostic Factors of Acute Kidney Injury
Brief Title: Etiology, Epidemiology and Prognostics of Acute Kidney Injury (AKI)
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Feng Ding,MD, professor, Huashan Hospital
Other Study IDs: KY2009-107
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Renal Failure; Nutrition Disorders
Keywords: acute kidney disease; prognosis; oxidative stress; inflammation; gene polymorphism
MeSH Terms: conditions — Renal Insufficiency; Nutrition Disorders; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1ml whole blood and 1ml serum will obtained within 24 hour after AKI for hematological and biochemistry analyze.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
* To investigate the etiology, epidemiology and prognostic factors of acute kidney injury.
* To find out risk factors that relate with the prognosis of acute kidney injury,focusing on inflammation, oxidative stress and nutritional status.
* To study on the relationship between gene polymorphism and prognosis of acute kidney injury.

DETAILED DESCRIPTION:
1. to investigate the relationship between preexisting malnutrition and adverse outcomes in patients with AKI

   - Several nutritional assessment methods such as anthropometric, clinical and biochemical evaluations have been used; however, no single indicator is considered to be a "gold standard."
2. to evaluate the association of serum nutritional variables and prognosis of acute kidney injury
3. Given the different half-lives of serum nutritional markers, we hypothesized that the utility of serum nutritional variables as prognostic predictors may differ in early death (<7 days) and late death (>7 days, <28 days) patients.

ELIGIBILITY:
Inclusion Criteria:

* age >=16 years and <= 88 years
* clinically diagnosed with acute kidney injury, according RIFLE or KDIGO criteria.

Exclusion Criteria:

* acute Renal Failure occurring in the setting of burns, obstructive uropathy, allergic interstitial nephritis, acute or rapidly progressive glomerulonephritis, vasculitis, hemolytic-uremic syndrome, thrombotic thrombocytopenic purpura (TTP), malignant hypertension, scleroderma renal crisis, atheroembolism, functional or surgical nephrectomy, hepatorenal syndrome, cyclosporin or tacrolimus nephrotoxicity
* Do Not Resuscitate (DNR) status
* subjects enrolled in another clinical trial that could affect the outcome of this study protocol

Ages: 16 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients selected from a university-affiliated hospital in Shanghai, China.
Sampling Method: Non-Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2009-04; Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
renal function survival rate days in the hospital days in the ICU | discharg from hospital, 28days,90days

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ding, professor, Principal Investigator — Huashan Hospital
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China

REFERENCES:
- [Derived] Gong Y, Ding F, Gu Y. Can Serum Nutritional Related Biomarkers Predict Mortality Of Critically Ill Older Patients With Acute Kidney Injury? Clin Interv Aging. 2019 Oct 18;14:1763-1769. doi: 10.2147/CIA.S218973. eCollection 2019. PMID 31695346
- [Derived] Yang T, Wang W, Tang X, Shi P, Zhang L, Yu W, Xie Y, Guo D, Ding F. Association between mineral and bone disorder in patients with acute kidney injury following cardiac surgery and adverse outcomes. BMC Nephrol. 2019 Oct 15;20(1):369. doi: 10.1186/s12882-019-1572-y. PMID 31615432
- [Derived] Gong Y, Ding F, Zhang F, Gu Y. Investigate predictive capacity of in-hospital mortality of four severity score systems on critically ill patients with acute kidney injury. J Investig Med. 2019 Dec;67(8):1103-1109. doi: 10.1136/jim-2019-001003. Epub 2019 Oct 1. PMID 31575668
- [Derived] Wang W, Hao G, Pan Y, Ma S, Yang T, Shi P, Zhu Q, Xie Y, Ma S, Zhang Q, Ruan H, Ding F. Serum indoxyl sulfate is associated with mortality in hospital-acquired acute kidney injury: a prospective cohort study. BMC Nephrol. 2019 Feb 14;20(1):57. doi: 10.1186/s12882-019-1238-9. PMID 30764800